CLINICAL TRIAL: NCT01686737
Title: Iyengar Yoga for Chemotherapy-induced Fatigue in Breast Cancer Patients
Acronym: IFaB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Postdoctoral fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012210
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Breast Neoplasms; Fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga (Experimental): Iyengar Yoga
  * 12 weeks of Iyengar yoga
  * 2 weekly sessions of 60 minutes
  Interventions: Behavioral: Iyengar Yoga
- Aerobic exercise (Active Comparator): Walking
  * 12 weeks of walking
  * 2 weekly sessions of 60 minutes
  Interventions: Behavioral: Walking
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Iyengar Yoga — * 12 weeks of Iyengar yoga
  * 2 weekly sessions of 60 minutes
  Arms: Yoga
Behavioral: Walking — * 12 weeks of walking
  * 2 weekly sessions of 60 minutes
  Arms: Aerobic exercise

SUMMARY:
Breast cancer is the most frequent cancer in women and is associated with profound restrictions of health-related quality of life and psychosocial health. More than three-quarters of women with breast cancer suffer from fatigue during cancer treatment. While exercise interventions can improve fatigue in breast cancer patients, many patients request complementary treatment approaches. Therefore, this study investigates the effects of yoga in women with breast cancer compared to aerobic exercise and usual care.

It is hypothesized that yoga is more effective than usual care and equally effective as aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* non-metastatic invasive breast cancer
* currently receiving adjuvant chemotherapy
* moderate to severe chemotherapy-induced fatigue
* physical and cognitive capacity to participate in yoga or walking

Exclusion Criteria:

* diagnosed and pharmacologically treated psychiatric disorder except depressive adaptation disorder as a reaction to cancer diagnosis
* ECOG status > 1
* prior malignancy with a disease-free survival < 10 years except curatively treated basalioma of the skin and carcinoma in situ of the cervix
* prior ductal carcinoma in situ (DCIS) ot the breast
* pregnancy or breastfeeding
* regular practice of yoga or walking during the past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Week 12
  Multidimensional Fatigue Inventory

SECONDARY OUTCOMES:
Fatigue | Week 36
  Multidimensional Fatigue Inventory
Health-related quality of life | Week 12, week 36
  Functional Assessment of Cancer Therapy - Breast
Depression and anxiety | Week 12, week 36
  Hospital Anxiety and Depression Scale
Sleep quality | Week 12, week 36
  Pittsburgh Sleep Quality Index
Perceived Stress | Week 12, week 36
  * Perceived Stress Scale
  * Impact of Event Scale
Salivary Cortisol | Week 12, week 36
  Cortisol awakening response
Safety | Week 0-36
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, PhD, Principal Investigator — University of Duisburg-Essen, Chair of Complementary and Integrative Medicine; Gustav J. Dobos, MD, Study Director — University of Duisburg-Essen, Chair of Complementary and Integrative Medicine
Locations (2):
- Germany (2):
  - Brustzentrum Köln-Hohenlind, St. Elisabeth-Krankenhaus Köln-Hohenlind, Cologne
  - Klinik für Senologie / Brustzentrum, Kliniken Essen-Mitte, Essen